CLINICAL TRIAL: NCT01185457
Title: Effect of Interscalene Block on Heart's Autonomic Nervous System With Heart Rate Variability Measurement
Brief Title: Effect of Interscalene Block on Heart Rate Variability (HRV)
Status: Completed | Type: Observational
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Eleni Chantzi, Anesthesiologist, Larissa University Hospital
Other Study IDs: HRVShoulder
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Shoulder Surgery; Beach Chair Position; Interscalene Block; HRV; Autonomic Nervous System
Keywords: Shoulder surgery; Beach chair position; Interscalene block; HRV; Autonomic nervous system

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Left interscalene block: Left shoulder surgery under left interscalene block and HRV
- Right interscalene block: Right shoulder surgery under right interscalene block and HRV

SUMMARY:
The Left interscalene block has a different effect on heart's autonomic nervous system, as measured with Heart Rate Variability, compared to Right interscalene block

ELIGIBILITY:
Inclusion Criteria:

* elective shoulder surgery
* Age 20- 45 years old
* ASA I - II

Exclusion Criteria:

* Coagulopathy disorders
* Infection at the puncture site for the interscalene block
* Neurologic deficit in the arm that is going to be operated
* Allergy to local anesthetics
* BMI > 35
* Psychiatric disorders
* Patient's refusal
* Problems with patient communication
* Arrythmia
* Ischaemic heart disease
* Diabetes mellitus
* Thyroid function disorders
* Patients with conduction disorders on the ECG
* Electrolyte disorders (K+, Na+, Ca++)
* Patients on medication that affect the ECG

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients for elective shoulder surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Effect of interscalene block on Heart Rate Variability (HRV) | 1 year
  The Left interscalene block has different effect on heart's autonomic nervous system, as measured with HRV, than the Right.

SECONDARY OUTCOMES:
Interscalene block and beach chair positioning | 2 years
  Effect of interscalene block on hypotension during beach chair positioning
Interscalene block and beach chair positioning | 2 years
  Effect of interscalene block on bradycardia during beach chair positioning

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Chantzi, Medicine, Principal Investigator — Larissa University Hospital; George Vretzakis, Medicine, Study Director — Larissa University Hospital; Metaxia Bareka, Medicine, Study Chair — Larissa University Hospital; Christos Iatrou, Medicine, Study Chair — Alexandroupoli University Hospital; Theophilos Karachalios, Medicine, Study Chair — Larissa University Hospital; Marina Simaioforidou, Medicine, Study Chair — Larissa University Hospital
Locations (1):
- Larissa University Hospital, Larissa, Thessaly, Greece

REFERENCES:
- [Background] Pomeranz B, Macaulay RJ, Caudill MA, Kutz I, Adam D, Gordon D, Kilborn KM, Barger AC, Shannon DC, Cohen RJ, et al. Assessment of autonomic function in humans by heart rate spectral analysis. Am J Physiol. 1985 Jan;248(1 Pt 2):H151-3. doi: 10.1152/ajpheart.1985.248.1.H151. PMID 3970172
- [Background] Pagani M, Lombardi F, Guzzetti S, Rimoldi O, Furlan R, Pizzinelli P, Sandrone G, Malfatto G, Dell'Orto S, Piccaluga E, et al. Power spectral analysis of heart rate and arterial pressure variabilities as a marker of sympatho-vagal interaction in man and conscious dog. Circ Res. 1986 Aug;59(2):178-93. doi: 10.1161/01.res.59.2.178. PMID 2874900
- [Background] Muzi M, Ebert Tj. Quantification of heart rate variability with power spectral analysis. Current Opinion in Aneasthesiology 6: 3-17, 1993
- [Background] Malliani A, Pagani M, Lombardi F, Cerutti S. Cardiovascular neural regulation explored in the frequency domain. Circulation. 1991 Aug;84(2):482-92. doi: 10.1161/01.cir.84.2.482. PMID 1860193
- [Background] RANDALL WC, ROHSE WG. The augmentor action of the sympathetic cardiac nerves. Circ Res. 1956 Jul;4(4):470-5. doi: 10.1161/01.res.4.4.470. No abstract available. PMID 13330193
- [Background] Rogers MC, Battit G, McPeek B, Todd D. Lateralization of sympathetic control of the human sinus node: ECG changes of stellate ganglion block. Anesthesiology. 1978 Feb;48(2):139-41. doi: 10.1097/00000542-197802000-00009. No abstract available. PMID 655444
- [Background] Schwartz PJ, Locati EH, Moss AJ, Crampton RS, Trazzi R, Ruberti U. Left cardiac sympathetic denervation in the therapy of congenital long QT syndrome. A worldwide report. Circulation. 1991 Aug;84(2):503-11. doi: 10.1161/01.cir.84.2.503. PMID 1860195